CLINICAL TRIAL: NCT00849316
Title: A Multicenter, Open Label, Nonrandomized, Non Interventional, Observational, Safety and Efficacy Study of NovoRapid™(Insulin Aspart) in Patients With Coexisting Diabetes and Kidney Disease in India. The NovoRapid™ Nephropathy Study
Brief Title: Safety and Efficacy Study of NovoRapid™ in Patients With Coexisting Diabetes and Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: Due to company decision to focus resources on the finalisation of three ongoing studies in the region
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-3702
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Safety and effectiveness data collection in connection with the use of the drug NovoRapid™ in patients with coexisting diabetes and chronic kidney disease in daily clinical practice.

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to investigate the clinical safety profile and effectiveness while using SC NovoRapid™ (insulin aspart) in patients with coexisting diabetes and kidney disease under normal clinical practice conditions in India.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with coexisting kidney disease and type 1 or type 2 diabetes is eligible for the study, including: newly-diagnosed subjects, insulin naïve and subjects who have received insulin or an insulin analogue before
* Subjects with kidney disease (stage I-IV) including transplant patients will be eligible for the study, if initiated with NovoRapid™"

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol requirements, e.g., uncooperative attitude, inability to return for the final visit
* Subjects with stage V of chronic kidney disease
* Subjects who previously enrolled in this study
* Known or suspected allergy to trial product(s) or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from both speciality practice settings who have been deemed appropriate to receive NovoRapid™ as new treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of major hypoglycaemic episodes | during 26 weeks

SECONDARY OUTCOMES:
Number of serious adverse events | during 26 weeks
Number of serious adverse drug reactions | during 26 weeks
Number of all daytime and nocturnal major hypoglycaemic events | during 26 weeks
Number of major hypoglycaemic events related to omission of a meal after injection | during 26 weeks
Number of all minor (daytime and nocturnal) hypoglycaemic events | during 4 weeks proceeding each study visits during Insulin Aspart (NovoRapidTM) therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Pathak, MD, Study Director — Novo Nordisk India Ltd; Ashok Moharana, MD, Study Director — Novo Nordisk India Private Ltd.

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com